CLINICAL TRIAL: NCT06251167
Title: A Multi-centre Feasibility Study Assessing Shoe-worn Insoles to Improve Clinical and Biomechanical Features of Knee Osteoarthritis
Brief Title: A Multi-centre Study of Shoe-worn Insoles and Knee Osteoarthritis
Acronym: MULTIWEDGE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Western University (Other); Dalhousie University (Other)
Responsible Party: Principal Investigator, Michael Hunt, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H22-03584
Record Dates: First submitted 2024-01-23; First posted 2024-02-09 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Orthotics; Foot pain; Biomechanics
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: We will conduct a two-arm, parallel group, multi-centre randomized controlled pilot study to assess the feasibility of our unique clinical biomechanics study, as well as the preliminary efficacy of the interventions on clinical and biomechanical outcomes at the feet and knees.
Who Masked: Participant, Investigator
Masking Description: Participants will be aware that there will be different types of insole interventions for this study, but will not be aware of the exact details of the insoles.
  Given that biomechanical assessment will be conducted in the intervention insole, it is not possible to mask the outcome assessor to intervention arm for participants. Instead, an investigator not involved in data collection will process all biomechanical data without knowledge of the intervention for a given participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lateral wedge insoles (LWIs) (Experimental): The LWIs will incorporate a 6 degree wedge along the lateral edge of the insole.
  Interventions: Device: Lateral wedge insoles (LWIs)
- Lateral wedge plus custom arch support (LWAS) (Experimental): The LWAS insoles will incorporate custom arch support along the medial edge as well as a 6 degree wedge along the lateral edge of the insole.
  Interventions: Device: Lateral wedge plus custom arch support (LWAS)

INTERVENTIONS:
Device: Lateral wedge insoles (LWIs) — Participants will be asked to wear these insoles in their own shoes for at least 5 hours per day for a period of 3 months. The LWIs will be constructed via 3D printing using a material of uniform density made to the length of the participant's feet, and will incorporate a 6 degree wedge along the lateral edge.
  Arms: Lateral wedge insoles (LWIs)
Device: Lateral wedge plus custom arch support (LWAS) — Participants will be asked to wear these insoles in their own shoes for at least 5 hours per day for a period of 3 months. These insoles will be designed based on an innovative tablet-based app designed by industry partner Kintec Footlabs, who will be the provider of the insoles for this project. Using the high-fidelity 3D scanning tool available (Apple's True Depth sensor), the Epitek Self-Scanner app captures tens of thousands of 3D data points within a single 1-second capture, and then uploads this foot data to a secure patient record system that is used for insole fabrication. The LWAS insoles will be comprised of variable density material (more dense laterally than medially) and milled directly to produce a full-length shell. The 6 degree wedge will be incorporated along the full lateral length of the insoles.
  Arms: Lateral wedge plus custom arch support (LWAS)

SUMMARY:
Shoe-worn insoles (also known as orthotics) can provide symptomatic relief for people with knee osteoarthritis. However, given they act at the feet, and given that many people with knee osteoarthritis also report foot pain, it is important to assess the effects of these devices at both joints. We will conduct a multi-centre randomized pilot trial to determine feasibility and preliminary efficacy.

ELIGIBILITY:
Inclusion Criteria:

* medial tibiofemoral OA defined as definitive osteophytes and joint space narrowing in the medial compartment, as confirmed with radiographs
* history of knee pain longer than 6 months
* average self-reported knee pain of at least 3 out of 10 (using an 11-point numerical rating scale with terminal descriptors of 0 = "no pain" and 10 = "worst pain imaginable") over the 6 months prior to baseline testing
* pain in the same foot/feet as the painful knee(s)
* ability to communicate in English
* show an immediate biomechanical response to the insoles. This final eligibility criterion will be determined from an in-person biomechanical assessment after participants have passed all previous eligibility screening.

Exclusion Criteria:

* radiographic evidence of more lateral tibiofemoral OA than medial
* knee surgery or intra-articular injection within the previous 6 months
* current or recent (within 6 months) corticosteroid use for any reason
* presence of a systemic arthritic condition
* history of knee joint replacement or tibial osteotomy
* any other condition affecting lower limb function
* current usage of shoe-worn insoles, or planning to acquire footwear modifications in the next 6 months
* any previous experience with insoles that resulted in increased lower limb pain or a self- or clinician-initiated termination of use.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment - number of screened patients who are eligible | from onset of recruitment through study completion
  The number of screened patients determined eligible to be enrolled in the study.
Retention - proportion of assessments with complete outcome measures data | immediately after the intervention
  Proportion of assessments with complete outcome measures data out of total number of assessments in the study protocol.
Insoles Delivery | from date of insoles ordering until date of delivery to the laboratory, assessed up to 3 months
  Time between foot scan assessment and delivery of insoles. Given that insoles will be manufactured centrally and distributed to the sites, we are interested in assessing the expected timeframe for enrollment in the study.
Self-reported knee pain | Baseline, 3 Months
  Knee pain will be measured by the Pain subscale (9 items) of the Knee Injury and Osteoarthritis Outcome Score (KOOS) at baseline and at 3-months. Each item is rated on a 5 points Likert scale where 0 = "No problems" and 4 = "Extreme Problems". Higher scores indicate better function. The scores are normalized to 0-100%.
Self-reported foot pain | Baseline, 3 Months
  Foot pain will be measured at baseline and at 3-months by the Pain subscale (7 items) of the Foot Function Index revised short form (FFI-RS). This is a self-report questionnaire consisting of 34 items that provides the ability to quantify aspects of foot pain, disability and activity limitation.
External knee adduction moment impulse | Baseline, 3 Months
  The external knee adduction moment impulse will be calculated. Participants will walk on an instrumented walkway (embedded force platform(s)) while high speed cameras track the trajectories of markers placed on bony landmarks. Moments will be calculated using an inverse dynamics approach.

SECONDARY OUTCOMES:
Self-reported overall physical function | Baseline, 3 Months
  Physical function will be measured by the Function, Daily Living subscale (17 items) of the Knee Injury and Osteoarthritis Outcome Score (KOOS) at baseline and at 3-months. Each item is rated on a 5 points Likert scale where 0 = "No problems" and 4 = "Extreme Problems". Higher scores indicate better function. The scores are normalized to 0-100%.
Self-reported foot function | Baseline, 3 Months
  Foot function will be measured at baseline and at 3-months by the Activity Limitations subscale (3 items) of the Foot Function Index revised short form (FFI-RS). This is a self-report questionnaire consisting of 34 items that provides the ability to quantify aspects of foot pain, disability and activity limitation.
External knee flexion moment impulse | Baseline, 3 Months
  The external knee flexion moment impulse will be calculated using the same methods as described for the external knee adduction moment impulse.
Self-selected gait speed | Baseline, 3 Months
  Self-selected gait speed will be calculated during the biomechanical gait analyses.
Rearfoot eversion peak | Baseline, 3 Months
  Participants will walk on an instrumented walkway while high speed cameras track the trajectories of markers placed on bony landmarks.

OTHER OUTCOMES:
Exit Interview | 3 months
  Participants will be invited to take part in semi-structured interviews, and asked about their knee and pain, their experiences with their insoles, and their attitudes towards different treatment approaches to manage knee OA. The purpose of this exploratory component will be to identify any themes related to the approach and design of the study that would need to be modified for the definitive RCT. Semi-structured interviews will be conducted to explore participants' attitudes and feelings about the interventions and the study design. The conversations will be recorded digitally, transcribed verbatim, and analyzed using a framework analysis. Themes will be developed, discussed, adjusted, and grouped in an iterative and inductive process. All data will be coded according to the final thematic index generated.

CONTACTS AND LOCATIONS:
Locations (1):
- Motion Analysis and Biofeedback Laboratory, Vancouver, British Columbia, Canada